CLINICAL TRIAL: NCT04365400
Title: A Randomised, Double-Blind, Placebo-Controlled, Dose Finding Phase IIb Study to Assess the Efficacy and Safety of Orally Administered Epeleuton in Patients With Hypertriglyceridemia and Type 2 Diabetes
Brief Title: Assess Efficacy and Safety of Epeleuton in Patients With Hypertriglyceridemia and Type 2 Diabetes
Acronym: TRIAGE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial prematurely terminated on 03 May 2022 due to the results from an interim analysis indicating a lack of efficacy in the study population.
Sponsor: Afimmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DS102A-07-CV1; 2020-000065-16 (EudraCT Number)
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Hypertriglyceridemia; Type 2 Diabetes
MeSH Terms: conditions — Hypertriglyceridemia; Diabetes Mellitus, Type 2 | interventions — epeleuton

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DS102 2000mg (Experimental): Participants in this group received 1000mg DS102 capsules twice daily.
  Interventions: Drug: DS102
- DS102 4000mg (Experimental): Participants in this group received 2000mg DS102 capsules twice daily.
  Interventions: Drug: DS102
- Placebo (Placebo Comparator): Participants in this group received placebo capsules twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DS102 — DS102 Epeleuton capsules
  Other Names: Epeleuton Capsules
  Arms: DS102 2000mg; DS102 4000mg
Drug: Placebo — Placebo capsules
  Other Names: Placebo Capsules
  Arms: Placebo

SUMMARY:
To assess the efficacy and safety of orally administered Epeleuton capsules versus placebo, in the treatment of adult patients with hypertriglyceridemia and type 2 diabetes

DETAILED DESCRIPTION:
This was a randomised, double-blind, Placebo-controlled, 3-arm, multi-centre Phase IIb study consisting of 26 weeks of active treatment and a 2-week post-treatment follow-up period in adult patients with hypertriglyceridemia and concomitant type 2 diabetes.

The screening period consisted of up to 6-weeks lead-in during which all patients were to undergo diet and lifestyle stabilisation, washout of disallowed medications and optimisation of statins.

After screening, patients were randomised (1:1:1) at the baseline visit into the following treatment groups:

* Treatment Group A (Placebo): four Placebo capsules orally administered twice a day, i.e., eight capsules daily for 26 weeks.
* Treatment Group B (Epeleuton 2g): two Epeleuton 500 mg capsules and two Placebo capsules orally administered twice a day, i.e., eight capsules daily for 26 weeks.
* Treatment Group C (Epeleuton 4g): four Epeleuton 500 mg capsules orally administered twice a day, i.e., eight capsules daily for 26 weeks.

The observation period was 32-34 weeks (lead-in: 4-6 weeks, treatment duration: 26 weeks, follow-up period: 2 weeks). During the study, 10 visits to the clinic were scheduled: two screening visits (Visit 1 and Visit 2), one visit at the start of the comparative treatment period (baseline/Visit 3), six visits in the comparative treatment period (Visit 4/Week 4, Visit 5/Week 8, Visit 6/Week 12, Visit 7/Week 16, Visit 8/Week 20 and Visit 9/Week 26 or Early Termination) and one final safety follow-up visit (Visit 10/Week 28).

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with type 2 diabetes mellitus at least 90 days prior to the first screening visit.
2. Patients with a HbA1C (glycosylated haemoglobin) between 7.0 - 10.0% (53-86 mmol/mol) (both inclusive)
3. Patients with a fasting triglyceride level ≥200 mg/dL (2.26 mmol/L) and <750mg/dL (8.46 mmol/L) at both screening visits.

   Note: If the triglyceride level is outside the required range at the second screening visit, an additional measurement can be obtained 1 week later, to confirm eligibility.

   Note: If a large difference in triglyceride level (>15%) is observed between screening 1 and screening 2, an additional measurement may be requested or patient may be deemed not eligible.
4. Patients who have been educated regarding diet and exercise at or before visit 1 (screening 1) and are willing to maintain and not alter a stable diet and activity routine throughout the study.
5. Patients who have been on a stable statin therapy at doses that are likely to achieve optimal LDL cholesterol and who are willing to continue this treatment throughout the study.

   Note: Stable statin therapy may consist of a statin with or without ezetimibe.
6. Patients with an LDL cholesterol level <130mg/dL (3.34 mmol/L) at both screening visits.
7. Patients who have a body mass index (BMI) ≥ 25kg/m2 and <50kg/m2.
8. Patients who have been on a stable daily dose of metformin (at least 1500mg or maximum tolerated dose for metformin monotherapy as documented in the subject medical record) and/or a sulfonylurea and/or a dipeptidyl peptidase-4 (DPP-4) inhibitor and/or a sodium-glucose transport protein 2 inhibitor (SGLT2i) and/or a GLP1-RA and/or basal insulin for at least 90 days prior to the day of first screening visit.

   Note: Dose of GLP1-RA must be stable for 6 months prior to baseline with no weight change >2kg for 3 months prior to baseline.

   Note: Dose of basal insulin must be stable for 4 months prior to baseline. All types of basal insulin are permitted, including insulin glargine, insulin degludec, insulin detemir, NPH insulin and pre-mixed insulin.
9. Female patients and male patients with female partners of childbearing potential must use highly effective contraceptive methods or have a sterilised partner for the duration of the study. Highly effective contraceptive methods are defined as methods that can achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include hormonal contraception, intrauterine device or sexual abstinence.

   Note: A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

   Note: Hormonal contraceptives must be on a stable dose for at least one month before baseline.

   Note: Sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient.
10. Patients whose pre-study or screening clinical laboratory findings do not interfere with their participation in the study, in the opinion of the Investigator, and do not violate any inclusion or exclusion criteria
11. Male or female patients aged 18 years and older on the day of signing the informed consent form (ICF).
12. Patients who are able to communicate well with the Investigator, to understand and comply with the requirements of the study, and understand and sign the written informed consent prior to initiation of any study specific activities or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Weissbach, MD, Study Director — Afimmune
Locations (56):
- United States (32):
  - US Site 5, Little Rock, Arkansas
  - US Site 23, Cerritos, California
  - US Site 18, Huntington Park, California
  - US Site 19, Los Angeles, California
  - US Site 20, Panorama City, California
  - US Site 21, Santa Ana, California
  - US Site 13, Santa Ana, California
  - US Site 15, Adairsville, Georgia
  - US Site 35, Ames, Iowa
  - US Site 2, Albany, New York
  - US Site 25, Hickory, North Carolina
  - US Site 11, Morehead City, North Carolina
  - US Site 34, Raleigh, North Carolina
  - US Site 26, Rocky Mount, North Carolina
  - US Site 28, Salisbury, North Carolina
  - US Site 32, Statesville, North Carolina
  - US Site 27, Wilmington, North Carolina
  - US Site 22, Edmond, Oklahoma
  - US Site 1, Wyomissing, Pennsylvania
  - US Site 3, Yardley, Pennsylvania
  - US Site 12, Jackson, Tennessee
  - US Site 7, Dallas, Texas
  - US Site 8, Fort Worth, Texas
  - US Site 14, Fort Worth, Texas
  - US Site 24, Houston, Texas
  - US Site 30, Houston, Texas
  - US Site 6, Houston, Texas
  - US Site 33, Houston, Texas
  - US Site 29, Missouri City, Texas
  - US Site 31, North Richland Hills, Texas
  - US Site 10, Waco, Texas
  - US Site 17, Winchester, Virginia
- Georgia (4):
  - Georgia Site 1, Batumi
  - Georgia Site 2, Kutaisi
  - Georgia Site 3, Kutaisi
  - Georgia Site 4, Tbilisi
- Germany (4):
  - Germany Site 7, Dresden
  - Germany Site 3, Hamburg
  - Germany Site 1, Heidelberg
  - Germany Site 5, Lübeck
- Israel (8):
  - Israel Site 9, Herzliya
  - Israel Site 1, Holon
  - Israel Site 5, Jerusalem
  - Israel Site 6, Jerusalem
  - Israel Site 4, Nahariya
  - Israel Site 8, Sakhnin
  - Israel Site 2, Tel Aviv
  - Israel Site 3, Tel Aviv
- Latvia (4):
  - Latvia Site 4, Ogre
  - Latvia Site 1, Riga
  - Latvia Site 2, Riga
  - Latvia Site 3, Riga
- Switzerland (4):
  - Switzerland Site 3, Lausanne
  - Switzerland Site 4, Lucerne
  - Switzerland Site 2, Olten
  - Switzerland Site 1, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 233 patients were randomized in a 1:1:1 ratio
Period: Overall Study
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
Started | 79 | 77 | 77
Completed | 49 | 50 | 50
Not Completed | 30 | 27 | 27

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: The SAS consists of all patients who received at least one dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo | Total
Number analyzed (Participants) | 79 | 77 | 77 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (9.3) | 58.9 (10.2) | 58.8 (10.1) | 59.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 28 | 92
  Male | 45 | 47 | 49 | 141
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 1 | 4
  White | 75 | 74 | 70 | 219
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Triglycerides From Baseline to Week 16
Description: Analysis of changes and percentage changes of triglycerides was performed using a Wilcoxon rank sum test with the Hodges Lehmann median and 95% confidence intervals estimates. For analysis of triglycerides, baseline was defined as the mean of the Baseline (Visit 3) and Screening 2/Week -1 (Visit 2) measurements.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS):
  Patients were included in the FAS, a modified intention-to-treat population, if they were randomised to the study, received at least one dose of study medication and had at least one post-baseline measurement.
Measure: Mean (Standard Error); unit: % Change in TG
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
Number analyzed (Participants) | 76 | 74 | 76
% Change in TG | -7.886 (4.096) | 5.273 (5.361) | -5.130 (4.945)
Statistical Analysis 1: Comparison: DS102 4000mg vs Placebo; Test type: Superiority; p = 0.1148124, Wilcoxon (Mann-Whitney); Hodges Lehmann Median = 8.24, 95% CI 2-sided [-2.01 to 18.19]
Statistical Analysis 2: Comparison: DS102 2000mg vs Placebo; Test type: Superiority; p = 0.8668467, Wilcoxon (Mann-Whitney); Hodges Lehmann Median = -0.82, 95% CI 2-sided [-10.16 to 7.96]

2. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Changes from baseline of HbA1c at each visit were analysed using mixed model analysis of covariance (ANCOVA) with baseline value as a covariate.
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % of HbA1c
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
Number analyzed (Participants) | 76 | 74 | 76
% of HbA1c | -2.255 (1.412) | -0.524 (1.162) | -0.503 (1.446)
Statistical Analysis 1: Comparison: DS102 4000mg vs Placebo; Test type: Superiority; p = 0.8658, ANCOVA; Difference in Change in HbA1c (%) = 0.02516, 95% CI 2-sided [-0.26658 to 0.316897]
Statistical Analysis 2: Comparison: DS102 2000mg vs Placebo; Test type: Superiority; p = 0.6500, ANCOVA; Difference in Change in HbA1c (%) = -0.07333, 95% CI 2-sided [-0.39012 to 0.243455]

3. Secondary Outcome: % Change in Triglycerides From Baseline to Weeks 4, 8, 12, 20 and 26
Description: Percent change in triglycerides from baseline to weeks 4, 8, 12, 20 and 26
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % Change in TG
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
Number analyzed (Participants) | 76 | 74 | 76
% Change in TG
  Week 4 - Baseline | -9.301 (3.994) | 5.965 (9.868) | -6.025 (4.479)
  Week 8 - Baseline | -5.018 (3.843) | -4.500 (4.623) | -5.242 (4.411)
  Week 12 - Baseline | -8.144 (4.071) | -4.215 (6.081) | 4.022 (5.532)
  Week 20 - Baseline | -5.666 (4.665) | 1.889 (5.005) | -4.270 (4.494)
  Week26 - Baseline | -8.213 (4.882) | 7.456 (6.585) | -0.675 (5.538)

4. Secondary Outcome: Change in HbA1c From Baseline to Weeks 4, 8, 12, 16 and 20
Description: Change in HbA1c (glycosylated haemoglobin) from baseline to weeks 4, 8, 12, 16 and 20
Time Frame: 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: % HbA1c
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
Number analyzed (Participants) | 76 | 74 | 76
% HbA1c
  Week 4 - Baseline | -2.606 (0.618) | -1.980 (0.683) | -1.365 (0.657)
  Week 8 - Baseline | -3.327 (0.978) | -2.933 (0.815) | -2.913 (0.861)
  Week 12 - Baseline | -3.448 (1.229) | -2.331 (1.052) | -1.315 (1.143)
  Week 16 - Baseline | -2.690 (1.338) | -1.733 (1.110) | -1.278 (1.216)
  Week 20 - Baseline | -4.176 (1.414) | -0.733 (1.188) | -0.811 (1.372)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Arm/Group | DS102 2000mg | DS102 4000mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 1/79 | 0/77 | 1/77
Other Adverse Events (participants affected / at risk) | 49/79 | 52/77 | 42/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS102 2000mg (N=79) | DS102 4000mg (N=77) | Placebo (N=77)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DS102 2000mg (N=79) | DS102 4000mg (N=77) | Placebo (N=77)
Diarrhoea (Gastrointestinal disorders) | 8 | 13 | 6
Nausea (Gastrointestinal disorders) | 2 | 6 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 2
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 1
Eructation (Gastrointestinal disorders) | 2 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 3 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Frequent Bowel Movements (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 7 | 2 | 5
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 0
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diarrhoea Infectious (Infections and infestations) | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Giardiasis (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1
Pulpitis Dental (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 4 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 4 | 0
Diabetes Melitus (Metabolism and nutrition disorders) | 1 | 0 | 2
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Taste Disorder (Nervous system disorders) | 1 | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 0 | 0 | 1
Depressed level of Consciousness (Nervous system disorders) | 0 | 0 | 1
Hypoesthesia (Nervous system disorders) | 1 | 0 | 0
Lacunar Stroke (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 2
Blood Triglycerides Increased (Investigations) | 1 | 0 | 1
Glomerular Filtration Rate Decreased (Investigations) | 0 | 2 | 0
Albumin Urine Present (Investigations) | 0 | 1 | 0
Blood Cholesterol Increased (Investigations) | 1 | 0 | 0
Blood Glucose Increased (Investigations) | 0 | 0 | 1
Blood Insulin Increased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1 | 0
Body Temperature Increased (Investigations) | 0 | 0 | 1
Electrocardiogram QRS Complex Abnormal (Investigations) | 0 | 1 | 0
Electrocardiogram T Wave Abnormal (Investigations) | 0 | 0 | 1
Glycosylated Haemoglobin Increased (Investigations) | 0 | 1 | 0
International Normalised Ratio Increased (Investigations) | 1 | 0 | 0
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0
Mean Cell Haemoglobin Concentration Decreased (Investigations) | 1 | 0 | 0
Mean Cell Haemoglobin Decreased (Investigations) | 1 | 0 | 0
Mean Cell Volume Decreased (Investigations) | 1 | 0 | 0
Occult Blood Positive (Investigations) | 1 | 0 | 0
QRS Axis Abnormal (Investigations) | 0 | 0 | 1
SARS-CoV-2 Test Positive (Investigations) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 1
Chest Pain (General disorders) | 2 | 0 | 0
Oedema Peripheral (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1
Hunger (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1
Vaccination Site Pain (General disorders) | 0 | 0 | 1
Atrioventricular Block First Degree (Cardiac disorders) | 0 | 1 | 1
Defect Conduction Intraventricular (Cardiac disorders) | 1 | 0 | 1
Bundle Branch Block Left (Cardiac disorders) | 0 | 1 | 0
Bundle Branch Block Right (Cardiac disorders) | 1 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1
Myocardial Failure (Cardiac disorders) | 1 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 5 | 0 | 3
Labile Hypertension (Vascular disorders) | 1 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 0 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Microalbuminuria (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Macule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Burns Third Degree (Injury, poisoning and procedural complications) | 0 | 1 | 0
Conjunctival Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 3 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0
Immunisation Reaction (Immune system disorders) | 0 | 0 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal Allergy (Immune system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1
Prostatic Dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1
Open Angle Glaucoma (Eye disorders) | 0 | 0 | 1
Vitreous Detachment (Eye disorders) | 1 | 0 | 0
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT04365400/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/00/NCT04365400/SAP_001.pdf